CLINICAL TRIAL: NCT03129087
Title: The Effect of Vocal Rest Versus Vocalization Following Xeomin® Injections in Spasmodic Dysphonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LawsonHRI2
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Adductor Spasmodic Dysphonia

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized, cross-over, clinical trial involving the comparison of two treatments (A and B) separated by a wash-out period (W). The patient participants will be randomized to one of the following two treatment orders: AWB or BWA.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vocal activity (Experimental): The vocal activity arm will require the participant to remain in the clinic and read aloud continuously for a period of one hour after a botulinum toxin injection
  Interventions: Behavioral: Vocal rest versus vocalization
- Vocal rest (Experimental): The vocal rest arm will require the participant to remain in the clinic and remain on complete vocal rest for a period of one hour after a botulinum toxin injection
  Interventions: Behavioral: Vocal rest versus vocalization

INTERVENTIONS:
Behavioral: Vocal rest versus vocalization — A comparison of one hour of vocal rest versus continuous vocalization after botulinum toxin injection

SUMMARY:
This study will compare the effects of vocal rest versus continuous vocalization for one hour immediately following botulinum toxin injections for adductor spasmodic dysphonia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adductor spasmodic dysphonia (ADSD) by an experienced neurologist and otolaryngologist. ADSD patients who have been stabilized on their treatment dose for at least 2 treatment cycles.

Exclusion Criteria:

* Diagnosed with another neurological disorder that is combined with ADSD (i.e. Parkinson's disease and ADSD). Previous history of an additional vocal pathology (i.e. vocal polps, vocal nodules, unilateral vocal fold paralysis, etc.)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Severity of spasmodic dysphonia symptoms | Six weeks post-treatment
  Acoustic measures and perceptual ratings of vocal spasm severity
Patient-reported outcome measures of symptoms and communication | six weeks post-treatment
  Six patient-reported questionnaires related to symptoms, communication effectiveness, quality of life, and self-efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- LawsonHRI, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No